CLINICAL TRIAL: NCT07338526
Title: Intensity Modulated PrOton Therapy in Pediatric BRain Tumors (IMPORT): A Phase 3 Randomized Controlled Trial
Brief Title: Intensity Modulated PrOton Therapy in Pediatric BRain Tumors (IMPORT)
Acronym: IMPORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tata Memorial Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4785
Record Dates: First submitted 2025-11-24; First posted 2026-01-14 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumor, Pediatric
Keywords: Brain tumor, Benign; Brain tumor, Pediatric
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, Phase 3 superiority, 2-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Other): Patients in the standard arm will undergo focal cranial radiotherapy using photons (X-rays) with Image Guided Intensity Modulated Radiotherapy(IG-IMRT) using Volumetric Modulated Arc Therapy(VMAT).
  Interventions: Radiation: Photon-based intensity-modulated radiation therapy (IMRT).
- Experimental Arm (Experimental): The patients in the experimental arm will undergo focal radiotherapy to an equivalent dose using protons with pencil beam scanning- IMPT or volumetric modulated proton arc therapy.
  Interventions: Radiation: Intensity-modulated proton therapy (IMPT)

INTERVENTIONS:
Radiation: Intensity-modulated proton therapy (IMPT) — Patients in the experimental arm will receive focal cranial radiotherapy using proton therapy delivered with IMPT or proton arc techniques. Dose prescriptions and volumes will match institutional standards independent of study allocation. Planning will include CT and MRI fusion, with target and OAR delineation identical to the control arm. Proton plans will use robust optimization and undergo multidisciplinary review. Treatment will be delivered with image guidance, with weekly toxicity monitoring and standard clinical and imaging follow-up.
  Arms: Experimental Arm
Radiation: Photon-based intensity-modulated radiation therapy (IMRT). — Patients in the control arm will receive focal cranial radiotherapy using photon-based IG-IMRT delivered with VMAT. Dose, fractionation, and target volumes will follow standard institutional protocols based on tumor type and molecular features. Planning CT and MRI fusion will guide contouring of GTV, CTV, PTV, and organs at risk. Treatment plans will be generated in the Treatment Planning System and reviewed in multidisciplinary meetings. Radiotherapy will be delivered on IGRT-equipped linear accelerators, with weekly assessments for acute toxicities and routine follow-up imaging as per standard care.
  Arms: Control Arm

SUMMARY:
Children diagnosed with benign or low-grade brain tumors often require radiation therapy to control their disease. While radiation can be effective, traditional techniques using X-rays (photon-based radiotherapy) expose healthy brain tissue to radiation, potentially leading to long-term side effects like memory loss, learning difficulties, hormone imbalances, hearing problems, and a higher risk of secondary cancers. This study, called the IMPORT Trial, aims to compare two types of radiation therapy-Intensity-Modulated Proton Therapy (IMPT) and Intensity-Modulated Radiation Therapy (IMRT)-to determine which is safer and more effective for children. IMPT, a newer technique, uses protons instead of X-rays to deliver radiation, reducing exposure to healthy brain tissue. Researchers believe this could help minimize long-term damage while maintaining effective tumor control.

What is the goal of the study?

The primary goal is to see if IMPT leads to better survival with fewer side effects compared to IMRT. The study will track how well children function over five years, looking at:

* Cognitive abilities (memory, attention, learning)
* Hormonal balance (pituitary gland function)
* Hearing ability
* Overall survival without significant decline in quality of life

How will the study work?

* Who can join? Children aged 6 to 16 years diagnosed with certain types of benign or low-grade brain tumors.
* How are patients treated? Patients will be randomly assigned to receive either IMRT or IMPT.
* What is analysed? Doctors will track survival, tumor control, cognitive function, endocrine health, and quality of life over time.
* How long will it take? The study will last 10 years (5 years to enroll patients, 5 years to follow up).

Proton therapy is more expensive and not widely available, so strong scientific evidence is needed to justify its use in routine treatment. If IMPT significantly improves quality of life and survival, it could become the preferred treatment, shaping future policies and making proton therapy more accessible for children who need it.

DETAILED DESCRIPTION:
Benign and low-grade primary brain tumors constitute a substantial proportion of pediatric central nervous system tumors and are associated with excellent long-term survival when managed with multimodality therapy. Despite favorable tumor control rates, survivors are at significant risk of treatment-related late effects, particularly following radiation therapy, which can adversely impact neurocognitive function, endocrine health, auditory function, and overall quality of life. Given the prolonged life expectancy of this population, minimizing radiation-induced toxicity while maintaining effective disease control is a major therapeutic priority.

Radiation therapy remains an essential curative modality for children with unresectable, residual, progressive, or recurrent benign and low-grade brain tumors. Advances in high-precision photon-based techniques such as intensity-modulated radiation therapy (IMRT) have improved dose conformality; however, photon therapy continues to expose large volumes of normal brain tissue to low and intermediate radiation doses. This exposure may lead to white matter injury, neuroinflammation, microvascular damage, and subsequent neurocognitive, endocrine, and auditory dysfunction, particularly in younger patients with developing brains.

Proton beam therapy offers a potential dosimetric advantage over photon therapy due to its physical depth-dose characteristics, allowing reduced integral dose to surrounding normal tissues. Intensity-modulated proton therapy (IMPT), delivered using pencil beam scanning, enables highly conformal dose distributions with improved sparing of organs at risk and may allow for reduction in treatment margins through enhanced image guidance and dose painting capabilities. These properties suggest a potential for meaningful reduction in late radiation-related toxicity in pediatric patients, while preserving tumor control.

While dosimetric and retrospective clinical data suggest advantages of proton therapy in reducing radiation exposure to critical neural structures, robust prospective randomized evidence demonstrating clinically meaningful benefits remains limited. Furthermore, the higher cost and limited availability of proton therapy necessitate careful evaluation of its value relative to advanced photon techniques, particularly in resource-constrained healthcare systems. Generating high-level evidence to guide patient selection and policy decisions is therefore essential.

The IMPORT trial is a prospective, randomized, open-label, phase III superiority study designed to compare IMPT with IMRT in children with benign and low-grade primary brain tumors treated with curative intent radiotherapy. The trial focuses on outcomes that are particularly relevant to long-term pediatric survivorship, including neurocognitive function, endocrine and auditory toxicity, and quality of life, while ensuring comparable tumor control.

The study introduces the concept of Qualified Overall Survival (qOS) as a composite primary endpoint that integrates survival, disease control, and clinically significant treatment-related morbidity. This composite endpoint is intended to capture outcomes that reflect both oncologic efficacy and functional preservation, thereby providing a patient-centered assessment of treatment benefit.

Participants will be randomized to receive either IMPT or IMRT, with radiation dose, fractionation, and target volumes determined by tumor type, location, and standard clinical practice. Tumor response and disease progression will be assessed using contemporary imaging-based criteria, while functional outcomes will be evaluated using standardized neurocognitive testing, endocrine assessments, audiological evaluations, and patient-reported quality-of-life instruments.

By directly comparing IMPT and IMRT in a randomized setting, the IMPORT trial aims to determine whether the dosimetric advantages of proton therapy translate into superior long-term functional outcomes and improved qualified survival, thereby informing evidence-based clinical decision-making and health policy for pediatric brain tumor management.

ELIGIBILITY:
Inclusion Criteria:

* Age at irradiation: 6 to 16 years
* Karnofsky/ Lansky Play Performance Status ≥ 60
* Diagnosis (histopathological/ radiological) of primary brain tumor with an expected survival of >5 years (e.g., circumscribed gliomas, low grade gliomas, low-grade glial/ glioneuronal tumors, meningioma, pituitary tumors, schwannoma, craniopharyngioma, ependymoma)
* Planned for focal cranial radiotherapy
* Informed consent taken

Exclusion Criteria:

* Re-irradiation
* Palliative radiotherapy
* Multifocal or multicentric disease
* Planned for whole brain irradiation or craniospinal irradiation
* Planned for hypo-fractionated or stereotactic radiotherapy

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 94 (Estimated)
Dates: Start 2025-08-07 (Actual); Primary Completion 2035-07-07 (Estimated); Study Completion 2035-07-07 (Estimated)

PRIMARY OUTCOMES:
Survival Outcome | 5 years
  Qualified Overall Survival (qOS) is a composite endpoint defined as survival without functional, cognitive, or quality-of-life deterioration, irrespective of whether the cause is disease progression or treatment toxicity. The study hypothesizes that IMPT is superior to IMRT for 5-year qOS. qOS is measured from randomization to the earliest of:
  1. death from any cause;
  2. radiological progression confirmed on multiparametric MRI with two scans ≥12 weeks apart or deemed progressive by multidisciplinary consensus;
  3. neurocognitive decline >10 IQ points on Wechsler scales;
  4. clinically significant hypopituitarism requiring hormonal supplementation (CTCAE v5 Grade ≥2);
  5. Grade ≥2 ototoxicity; or
  6. symptomatic radiation necrosis requiring corticosteroids >4 weeks or anti-angiogenic therapy (e.g., bevacizumab).

SECONDARY OUTCOMES:
Overall Survival (OS) | At 5 years
  Overall Survival (defined as the time elapsed between date of randomisation to death due to any cause)
Progression-free Survival (PFS) | at 5 years
  Progression-free survival(defined as the time elapsed between date of randomisation to documented clinico-radiological progression or death)
Quality of Life indices | Pre-Radiotherapy (Baseline), Radiotherapy conclusion- within 1 week, 3-months post RT, 1-year post RT, annually till 5-years
  Quality of life assessed using patient-reported outcome measures developed by the European Organisation for Research and Treatment of Cancer (EORTC), including the core and disease-specific modules administered in this study. Scores are linearly transformed to a range of 0 to 100. For functional scales and global health status, higher scores indicate better quality of life; for symptom scales, higher scores indicate worse symptoms. Assessed at baseline and follow-up.
  Unit of Measure: Units on a scale
Cost-effectiveness based on EQ-5D-5L derived utilities | Pre-Radiotherapy (Baseline), Radiotherapy conclusion- within 1 week, 3-months post RT, 1-year post RT, annually till 5-years
  Health-related quality of life for economic evaluation will be assessed using the EuroQol 5-Level 5-Dimension questionnaire (EQ-5D-5L). Responses will be converted to utility scores using a country-specific value set and used to estimate quality-adjusted life years (QALYs) for cost-effectiveness analysis. Assessed at baseline and follow-up.
  Unit of Measure: Quality-adjusted life years (QALYs)
Response Rate (RR) | Radiotherapy conclusion- within 1 week, 3-months post RT, 1-year post RT, annually till 5-years
  Response Rate (complete and partial response) as decided by contemporary image-based response criteria (RAPNO, RANO-LGG 2.0)
Sub-domain of qOS | Radiotherapy conclusion- within 1 week, 3-months post RT, 1-year post RT, annually till 5-years
  Cumulative incidence of sub-domains of qualified overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Tata Memorial Hospital, Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: No